CLINICAL TRIAL: NCT06425263
Title: Microfragmented Adipose Tissue Injection Compared to Hyaluronic Acid for Treatment of Temporomandibular Joint Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mutaz Alkhair Hamad Elsayed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMFS 335
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Temporomandibular Joint Osteoarthritis

STUDY DESIGN:
Intervention Model Description: comparison between injection of hyaluronic acids and adipose tissue in temporomandibular joint
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injection with adipose tissue (Experimental): After standard arthrocentesis of the temporomandibular joint
  * Direct access to the buccal fat pad, is found at distobuccal depth of the maxillary tuberosity.
  * It may be dissected during the resection an upper mucosal incision posterior to the second molar
  * After a single scissor stab through the periosteum the (BFP)extrude into the operative site.
  * Closure of the flap by suitable suture.
  * Collection of lipids then manually manipulated with two syringes connecting together and pushing the lipids against each other to receive the injectable amount of micro fragmented adipose tissue .
  Interventions: Biological: adipose tissue fragmented
- injection with hyaluronic acids (Active Comparator): Arthrocentesis of the superior joint compartment was performed in all patients under local anesthesia using the technique described by Nitzan et al.
  Another 19-gauge needle was inserted into the distended compartment in the area of the articular eminence, and the superior joint space was irrigated with 200 mL saline solution, allowing a free flow through the first needle.
  On termination of procedure, 2 mL commercially available hyaluronic injected into the superior compartment.
  Interventions: Biological: adipose tissue fragmented

INTERVENTIONS:
Biological: adipose tissue fragmented — harvested from the case form buccal pad of fat

SUMMARY:
Internal derangement and osteoarthritis are the most common degenerative temporomandibular joint diseases and initial treatment for such conditions relies on arthrocentesis.

Micro fragmentation of adipose tissue has been proven in orthopedic literature to represent a more effective method to preserve stem cells, but no application has ever been reported in the temporomandibular joint.

DETAILED DESCRIPTION:
Rationale for conducting the research:

The rationale of this procedure is to remove inflammatory mediators, reduce friction, stimulate the production of new synovial fluid, eliminate suction-cup effect.

The purpose of this study was to evaluate the hypothesis that TMJ arthrocentesis with intraarticular injection of autologous micro fragmented adipose tissue leads to better clinical outcomes in terms of reducing pain and improving function

compared with arthrocentesis and intraarticular injection of hyaluronic acid (HA) in patients with TMJ internal derangement and osteoarthritis.

Preliminary results of this clinical trial show that the injection of micro fragmented adipose tissue can significantly improve outcomes of pain and function compared with the standard treatment and encourage to pursue research on this topic.

Further studies with a longer follow-up time are needed to evaluate the clinical stability of the achieved improvement in pain and function.

For this reason, this protocol has been designed with the aim to investigate whether injection in the TMJ of micro fragmented fat tissue can achieve the same improvements of pain and function, compare this technique with standard arthrocentesis with HA injection.

ELIGIBILITY:
Inclusion Criteria:

* * TMJ osteoarthritis assessed by clinical examination and MRI imaging

  * Presence of TMJ-related symptoms including at least limited mouth opening and joint pain
  * Previously failed conservative treatment
  * Age superior to 14 years
  * No previous TMJ surgical procedures
  * Acquisition of informed consent;
  * Complete availability of the data acquired preoperatively and during each follow-up
  * Patients free from any systemic disease that may affect the procedure.

Exclusion Criteria:

* * Previously diagnosed hematological and neurological conditions;

  * Previous malignant head and neck neoplasms;
  * Contraindication to fat harvesting.
  * Uncooperative patients.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — age superior to 14 years of age
Enrollment: 28 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
VAS | 3 months
  by Vas measurement scale OF PAIN

SECONDARY OUTCOMES:
mouth opening | 3 months
  degree of opening on each visit

IPD SHARING:
Plan to Share IPD: Yes
Dose Lipogems injection affect TMJ derangement more than hyaluronic acid in treatment of the temporomandibular joint osteoarthritis and internal derangement?
  Statement of the problem:
  Internal derangement and osteoarthritis are the most common degenerative temporomandibular joint diseases and initial treatment for such conditions relies on arthrocentesis.
  Micro fragmentation of adipose tissue has been proven in orthopedic literature to represent a more effective method to preserve stem cells, but no application has ever been reported in the temporomandibular joint.
Supporting Information: CSR
Time Frame: WITH IN THIS YEAR